CLINICAL TRIAL: NCT03056274
Title: METformin in Intrahepatic Cholestasis of Pregnancy (METRIC) Study
Brief Title: Metformin in Intrahepatic Cholestasis of Pregnancy
Acronym: METRIC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Epsom and St Helier University Hospitals NHS Trust (Other)
Collaborators: King's College Hospital NHS Trust (Other); Medway NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RVR
Record Dates: First submitted 2016-12-22; First posted 2017-02-17 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-01

CONDITIONS: Intrahepatic Cholestases; Pregnancy Complications
Keywords: Metformin; Ursodeoxycholic acid; Outcomes
MeSH Terms: conditions — Cholestasis, Intrahepatic; Pregnancy Complications | interventions — Metformin; Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin arm (Active Comparator): Metformin
  Interventions: Drug: Ursodeoxycholic Acid
- Ursodeoxycholic acid (Active Comparator): Ursodeoxycholic acid
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin Hydrochloride (HCl) Tablets, is an oral antihyperglycemic drug used in the management of type 2 diabetes
  Other Names: Glucophage
  Arms: Ursodeoxycholic acid
Drug: Ursodeoxycholic Acid — Ursodeoxycholic acid (UDCA) is used to treat gallstones and primary biliary cirrhosis. UDCA is also used to treat obstetric cholestasis (OC), a liver condition that occurs specifically in pregnancy.
  Other Names: Destolit®, Urdox®, Ursofalk®, Ursogal®
  Arms: Metformin arm

SUMMARY:
This is a pilot study aimed at comparing the effect of metformin versus ursodeoxycholic acid in women with intrahepatic cholestasis in pregnancy. The study will be conducted in three NHS hospital sites, over an 18 month period.

DETAILED DESCRIPTION:
Intrahepatic cholestasis is a condition that affects pregnant women. It is characterised by itching, usually in the third trimester of pregnancy and is associated with an increase in the liver enzymes and bile salts. This can be associated with maternal and neonatal morbidity, and rarely perinatal mortality.

The investigators propose to assess and compare the effect of Metformin versus Ursodeoxycholic acid on lowering liver enzymes and bile salts, improving maternal morbidity and improving neonatal outcomes.

This study is a pilot study that will be conducted at 3 NHS hospital sites where patients will randomly assigned to receive either Metformin or Ursodeoxycholic acid. There will be 20 patient in each arm. Recruitment will commence in February 2017 and will run for an 18 month period.

ELIGIBILITY:
Inclusion Criteria:

1. 20+0 to 40 weeks' gestation on day of randomisation
2. Itching with a raised serum bile acid above the upper limit of normal
3. Normal anomaly scan at 20 weeks
4. Aged 18 years or over
5. Able to give written informed consent
6. No known pre-existing liver disease

Exclusion Criteria:

1. Decision already made for delivery within the next 48 hours
2. Known allergy to any component of the ursodeoxycholic acid or metformin tablets
3. Patients already on metformin for other conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Normalisation of maternal serum concentration of bile salts and liver enzymes | From date of randomisation to date of delivery assessed up to 26 weeks
  Normalisation of Bile acids and liver enzymes - both parameters are the cornerstone for a diagnosis of intrahepatic cholestasis. They have been separated into two outcomes due to to the different laboratory indices of measurement. Results will be aggregated together to report number of patients with abnormal results
Normalisation of maternal serum concentration of liver enzymes | From date of randomisation to date of delivery assessed up to 26 weeks
  Normalisation of liver enzymes Alanine transaminase Aspartate transaminase Bilirubin (total) Gamma glutamyl transferase Results will be aggregated together to report the number of patients with abnormal liver enzymes

SECONDARY OUTCOMES:
Fetal outcomes | From date of randomisation to date of delivery assessed up to 26 weeks
  Perinatal death
Fetal outcomes | From date of randomisation to date of delivery assessed up to 26 weeks
  Preterm delivery
Fetal outcomes | Immediately upon delivery date
  Respiratory distress syndrome
Fetal outcomes | Immediately upon delivery date
  Birth weight (g)
Fetal outcomes | Immediately upon delivery date
  Birth weight percentile
Fetal outcomes | Immediately upon delivery date
  Gestational age at delivery

OTHER OUTCOMES:
Fetal outcomes | Immediately upon delivery date
  Presence of meconium
Fetal outcomes | Immediately upon delivery date
  APGAR score at 5 minutes
Fetal outcomes | Immediately upon delivery date
  Umbilical arterial pH at birth
Maternal outcomes | From date of randomisation to date of delivery assessed up to 26 weeks
  Symptoms (itch) - assessed by questionnaire at clinic visits
Maternal outcomes | From date of randomisation to date of delivery assessed up to 20 weeks
  Maximum dose of medication required
Maternal outcomes | From date of randomisation to date of delivery assessed up to 20 weeks
  Gestational diabetes
Maternal outcomes | From date of randomisation to date of delivery assessed up to 26 weeks
  Postpartum haemorrhage
Maternal outcomes | From date of randomisation to date of delivery assessed up to 20 weeks
  Mode of delivery
Maternal outcomes | From date of randomisation to date of delivery assessed up to 26 weeks
  Liver failure

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Shehata, FRCPI, FRCOG, Principal Investigator — Epsom & St Helier University Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elfituri A, Ali A, Shehata H. Managing Recurring Obstetric Cholestasis With Metformin. Obstet Gynecol. 2016 Dec;128(6):1320-1323. doi: 10.1097/AOG.0000000000001748. PMID 27824743
- [Derived] Walker KF, Chappell LC, Hague WM, Middleton P, Thornton JG. Pharmacological interventions for treating intrahepatic cholestasis of pregnancy. Cochrane Database Syst Rev. 2020 Jul 27;7(7):CD000493. doi: 10.1002/14651858.CD000493.pub3. PMID 32716060